CLINICAL TRIAL: NCT03504605
Title: The Role of Parental Perfectionistic Cognitions in an Intervention to Improve Self- Compassion and Reduce Shame: Findings in the Context of Child Chronic Health Conditions
Brief Title: Impact of Parental Perfectionistic Cognitions Self-compassion Intervention Effects on Shame in Child Health Context
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sheffield (Other)
Collaborators: Sheffield Children's NHS Foundation Trust (Other); Alder Hey Children's NHS Foundation Trust (Other); Chesterfield Royal NHS Foundation Trust (Unknown)
Responsible Party: Principal Investigator, Catherine Lilley, Principal Investigator, University of Sheffield
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 155657
Record Dates: First submitted 2018-04-06; First posted 2018-04-20 (Actual); Last update posted 2019-07-26 (Actual); Status verified 2019-07

CONDITIONS: Diabetes Mellitus, Type 1; Epilepsy; Asthma; Shame; Self-Compassion; Stress; Perfectionistic Cognitions
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Epilepsy; Asthma

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-compassion intervention (Experimental): Participants will be asked to recall and write (in an online text-box) about a parenting event during which they felt shame. They will then receive the online self-compassion intervention as detailed in Sirois, Bögels and Emerson (in revision). This involves parents in the experimental condition being given a validated set of instructions asking them to reflect on the event and write self-compassionate responses (see intervention).
  Interventions: Other: Online self-compassion intervention
- Control (No Intervention): Participants will be asked to recall and write (in an online text-box) about a parenting event during which they felt shame. Those in the control condition will be asked to re-read the account of the event and make notes about factual information (e.g. time of day, who was there, etc.). It should be noted that if the SCI is found to reduce state shame and increase state self-compassion, it will be offered to participants in the control group.

INTERVENTIONS:
Other: Online self-compassion intervention — Parents are asked to write in an online text box about a parenting event in which they felt shame. They are then given a validated set of instructions asking them to reflect on the event and write self-compassionate responses.
  Arms: Self-compassion intervention

SUMMARY:
Parents of children with long-term health conditions (LTCs) can experience shame related to parenting. Whilst self-compassion interventions (SCIs) can reduce parental shame, this has not been studied with parents of children with LTCs. Perfectionistic cognitions may also moderate the effects of SCIs. This study will test an online SCI with parents of children with type 1 diabetes, epilepsy or asthma. Parents will complete online questionnaires pre- and post a SCI/control intervention. Hypotheses will be tested using analysis of covariance and moderation analysis. Findings will enhance knowledge of vulnerability factors to distress for parents of children with LTCs, and inform interventions.

DETAILED DESCRIPTION:
This study is part of a joint project being conducted in the University of Sheffield by another Trainee Clinical Psychologist. The studies use the same baseline, but only this study includes a clinical trial.

Parents of children with long-term health conditions (LTCs) can experience shame related to parenting. Whilst self-compassion interventions (SCIs) have been shown to reduce parental shame, this has not been studied with parents of children with LTCs. Evidence also suggests that perfectionistic cognitions may moderate the effects of SCIs. This study will test an online SCI with parents of children with type 1 diabetes, epilepsy or asthma.

This design of the study is experimental and prospective. The methodology is made up of two parts:

1. Baseline data collection period:

   Baseline measures of perfectionistic cognitions, state and trait self-compassion, state shame and parental stress relating to their child's LTC will be taken, alongside demographic information regarding the participant's age, gender, their child's type of LTC and duration of illness (which research indicates affects levels of self-compassion or perfectionistic cognitions).

   At baseline, all participants will also be asked to give their email contact details. Qualtrics will be set up to randomise participants' emails into one of two groups at baseline so that participants can be allocated to one of the follow-up studies.
2. Follow-up experimental study:

Eligible participants will be randomised (as described above) into this experimental follow-up study or that of the other Trainee Clinical Psychologist. On entry to this study they will be further randomised via Qualtrics into an experimental (self-compassion intervention) or control group.

Both groups will be asked to recall and write (in an online text-box) about a parenting event during which they felt shame. Those in the experimental group will receive the online self-compassion intervention as detailed in Sirois, Bögels and Emerson (in revision). This involves parents in the experimental condition being given a validated set of instructions asking them to reflect on the event and write self-compassionate responses. Participants in the control condition will be asked to re-read the account of the event and make notes about factual information (e.g. time of day, who was there, etc.).

Measures of state and trait self-compassion, shame and parental stress related to their child's LTC will be repeated immediately after the intervention. The parent will then complete a mood neutralisation task (requiring them to write about a time that they felt proud of their parenting). Parents randomised to the control condition will receive the self-compassion intervention retrospectively, if results indicate it was effective.

Hypotheses:

1. Parents of children with a chronic health condition will report reduced state shame associated with parenting after the self-compassion intervention, compared with those in the control condition.
2. Parents of children with a chronic health condition will report an increase in state self-compassion after the self-compassion intervention, compared with those in the control condition.
3. High levels of shame will relate to lower self-esteem and higher perfectionistic cognitions, with a relationship present over time.
4. The intervention will be less effective for those high in perfectionistic cognitions (i.e. will be moderated by parents' levels of PCs).

ELIGIBILITY:
Inclusion Criteria:

* Parents (mothers and fathers, biological or non-biological) with a child under 18 years and living with them)
* Parents with children with a medical diagnosis of Type 1 diabetes mellitus, asthma, or epilepsy.

Exclusion Criteria:

* Parents and / or children who are currently receiving or who have engaged in therapy for stress related issues, with regards to the child's diagnosis.
* Parents who don't have access to a computer.
* Parents who have difficulties with reading.
* Parents who aren't fluent in English.

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 344 (Actual)
Dates: Start 2018-08-15 (Actual); Primary Completion 2019-01-23 (Actual); Study Completion 2019-07-25 (Actual)

PRIMARY OUTCOMES:
Self-compassion Scale | Change from baseline trait self-compassion through to study completion (anticipated one week).
  Outcome measure to assess trait self-compassion, which is defined as a trait in which people are mindful to emotions and respond towards themself with kindness and with a sense of common humanity, through difficulties, or following perceived failure/ personal shortcomings
PANAS-X | Change from baseline shame through to study completion (anticipated one week).
  Outcome measure to assess shame, defined as a self-conscious emotion, distinct from guilt as it is constructed of negative evaluation directed towards the self (as opposed to behaviours).
Self-compassion items | Change from baseline state self-compassion through to study completion (anticipated one week).
  An adapted outcome measure to assess state self-compassion, defined as self-compassion that can change in the moment.

OTHER OUTCOMES:
Perfectionistic cognitions Inventory | Change from baseline perfectionistic cognitions through to study completion (anticipated one week).
  Outcome measure to assess automatic perfectionistic thoughts, defined as automatic thoughts to do with perfection. They are included in this study as potential moderator of the impact of the intervention on shame and self-compassion.
Pediatric Inventory for Parents | Change from baseline parental stress through to study completion (anticipated one week).
  Outcome measure to assess parental stress

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Lilley, Principal Investigator — University of Sheffield; Georgina Rowse, Study Director — University of Sheffield; Fuschia Sirois, Study Director — University of Sheffield; Amrit Sinha, Study Director — University of Sheffield; Kirsteen Meheran, Principal Investigator — University of Sheffield
Locations (1):
- Sheffield Childrens Hospital, Sheffield, United Kingdom

IPD SHARING:
Plan to Share IPD: No